CLINICAL TRIAL: NCT01981603
Title: Transplant Navigator Dissemination
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Catherine Sullivan (Other)
Responsible Party: Sponsor-Investigator, Catherine Sullivan, Center Manager, Research, MetroHealth Medical Center
Organization: MetroHealth Medical Center (Other)
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: IRB12-00660
Record Dates: First submitted 2013-10-30; First posted 2013-11-11 (Estimated); Last update posted 2018-03-22 (Actual); Status verified 2018-03

CONDITIONS: Kidney Transplant; Renal Failure Chronic Requiring Hemodialysis
Keywords: Navigators; Kidney Transplant; Hemodialysis

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- navigator (Experimental): Kidney transplant recipients will serve as navigators to educate and assist other patients with the transplant process.
  Interventions: Other: navigator
- usual care (No Intervention): usual care

INTERVENTIONS:
Other: navigator
  Arms: navigator

SUMMARY:
Primary Aim A. To disseminate and determine the impact of streamlined navigation on wait listing and number of transplants. The navigator will provide tailored information and assistance to help dialysis patients complete the tasks required at each step in the transplant process. In the control group, dialysis patients will continue to get usual care from their nephrologists and dialysis facility personnel.

Hypothesis: Compared to control patients, intervention patients will be significantly more likely to be wait listed or receive a kidney transplant.

ELIGIBILITY:
Inclusion Criteria:

* between the ages of 18-70
* receiving in center hemodialysis

Exclusion Criteria:

* less than 18 years of age
* older than 70 years of age

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1926 (Actual)
Dates: Start 2014-01-01 (Actual); Primary Completion 2017-12 (Actual); Study Completion 2017-12 (Actual)

PRIMARY OUTCOMES:
The proportion of patients who are wait listed or receive a kidney transplant. | approximately 3 years

CONTACTS AND LOCATIONS:
Locations (5):
- United States (5):
  - Lutheran Hospital, Fort Wayne, Indiana
  - University of Kentucky, Lexington, Kentucky
  - Jewish Hospital, Louisville, Kentucky
  - MetroHealth Medical Center, Cleveland, Ohio
  - The Ohio State University, Columbus, Ohio